CLINICAL TRIAL: NCT04316403
Title: Evaluation of the Efficacy of Laser-assisted Flapless Corticotomy in Accelerating Canine Retraction: A Split-mouth Randomized Controlled Clinical Trial
Brief Title: Laser-assisted Flapless Corticotomy in Accelerating Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-01-2020
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Class II Division 1 Malocclusion; Maxillary Prognathism; Protrusion, Incisor
Keywords: Tooth movement; Acceleration of tooth movement; Er:YAG laser-assisted corticotomy
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-assisted corticotomy (Experimental): Er:YAG laser beam was used to perform several perforations to the alveolar bone around the canine in one side of the mouth hoping that would accelerate canine retraction
  Interventions: Procedure: Er:YAG laser
- Traditional treatment (No Intervention): Canines in this group were retracted by the conventional manner.

INTERVENTIONS:
Procedure: Er:YAG laser — This application was made before the onset of canine retraction in one side of the mouth
  Arms: Laser-assisted corticotomy

SUMMARY:
Erbium lasers have been suggested to accomplish corticotomy without flap reflection due to their attractive advantages. The current trial aimed to evaluate the efficacy of laser-assisted flapless corticotomy in accelerating orthodontic tooth movement. The secondary aim was to evaluate the patients' responses to laser application. It was postulated that canine retraction after laser-assisted flapless corticotomy would be accomplished within a shorter period compared with the conventional canine retraction method, with no significant degree of pain and discomfort.

DETAILED DESCRIPTION:
Comprehensive orthodontic treatment with fixed appliances usually takes more than 18 months in mild and severe cases. Prolonged treatment time can cause many adverse effects such as pain, discomfort, external root resorption, white spots and dental caries. Decreasing the treatment time for tooth movement has been the focus of both the clinicians and the patients. For the last few decades, investigators have recommended many treatment approaches intending to reduce overall treatment time such as low friction and self-ligating bracket systems, low-level laser irradiation, electrical currents, pharmacological approaches, local platelet-rich plasma (PRP) injection and surgical approaches like dentoalveolar distraction and selective alveolar decortication or corticotomy

ELIGIBILITY:
Inclusion Criteria:

* Class II division 1 patients requiring orthodontic treatment with fixed appliances and a need for upper first-premolar extraction using a two-step retraction technique.
* Permanent dentition with an age range from 16 to 24 years.
* Healthy with no systemic conditions.
* Adequate oral hygiene and healthy periodontal tissues
* no previous orthodontic treatment
* Absence of canine endodontic treatment.

Exclusion Criteria:

* Bimaxillary dentoalveolar severe protrusion.
* Previous orthodontic treatment.
* Subject with psychological abnormalities.
* Subject with systemic diseases.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Change in the canine retraction rate | 10 minutes after laser application, one, two, four, 8 and 12 weeks after laser application
  The distance between the first molar labial hook and the canine bracket hook was recorded using Digital Boely gauge and then this distance was divided by the time that passed between two assessment points.

SECONDARY OUTCOMES:
Change in the levels of pain and discomfort | at the 1st day following laser application (10 minutes) and at the 3rd, 5th and 7th days following laser application
  A questionnaire was administered at the 1st, 3rd, 5th and 7th day after laser application. The questionnaire contained 5 questions (using 4-point Likert ordinal scales) to collect patients' responses on the following questions:
  Question 1: Do you feel pain during eating? Question 2: Do you feel pain during the day? Question 3: Do you feel pain that can awaken you during the night? Question 4: Do you feel swollen on the surgical side?
  The possible answers were:
  1. No 2.Mild 3.Moderate 4. Severe For the first four questions, the higher the score, the worse the feeling was.
  Question 5: Which one of the following has caused more discomfort to you?
  1. Extraction of premolars 2. Laser application 3.Both

CONTACTS AND LOCATIONS:
Overall Officials: Samer T Jaber, DDS MSc, Principal Investigator — PhD student, Orthodontics Department, University of Damascus Dental School; Rabab Al-sabbagh, DDS MSc PhD, Study Chair — Professor of Orthodontics, University of Hama, Hama, Syria
Locations (1):
- Orthodontic Department, University of Hama Dental School, Hama, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher MA, Wenger RM, Hans MG. Pretreatment characteristics associated with orthodontic treatment duration. Am J Orthod Dentofacial Orthop. 2010 Feb;137(2):178-86. doi: 10.1016/j.ajodo.2008.09.028. PMID 20152672
- [Background] Segal GR, Schiffman PH, Tuncay OC. Meta analysis of the treatment-related factors of external apical root resorption. Orthod Craniofac Res. 2004 May;7(2):71-8. doi: 10.1111/j.1601-6343.2004.00286.x. PMID 15180086
- [Background] Uribe F, Padala S, Allareddy V, Nanda R. Patients', parents', and orthodontists' perceptions of the need for and costs of additional procedures to reduce treatment time. Am J Orthod Dentofacial Orthop. 2014 Apr;145(4 Suppl):S65-73. doi: 10.1016/j.ajodo.2013.12.015. PMID 24680026
- [Background] Hassan SE, Hajeer MY, Alali OH, Kaddah AS. The Effect of Using Self-ligating Brackets on Maxillary Canine Retraction: A Split-mouth Design Randomized Controlled Trial. J Contemp Dent Pract. 2016 Jun 1;17(6):496-503. doi: 10.5005/jp-journals-10024-1879. PMID 27484605
- [Background] AlSayed Hasan MMA, Sultan K, Hamadah O. Low-level laser therapy effectiveness in accelerating orthodontic tooth movement: A randomized controlled clinical trial. Angle Orthod. 2017 Jul;87(4):499-504. doi: 10.2319/062716-503.1. Epub 2016 Nov 21. PMID 27869476
- [Background] Hashimoto H. Effect of micro-pulsed electricity on experimental tooth movement. Nihon Kyosei Shika Gakkai Zasshi. 1990 Aug;49(4):352-61. PMID 2133892
- [Derived] Jaber ST, Al-Sabbagh R, Hajeer MY. Evaluation of the efficacy of laser-assisted flapless corticotomy in accelerating canine retraction: a split-mouth randomized controlled clinical trial. Oral Maxillofac Surg. 2022 Mar;26(1):81-89. doi: 10.1007/s10006-021-00963-x. Epub 2021 Apr 20. PMID 33876339